CLINICAL TRIAL: NCT01369095
Title: A Multicenter, Randomized, Double-Blind, Active Controlled, Comparative, Fixed-Dose, Dose Response Study of the Efficacy and Safety of BMS-820836 in Patients With Treatment Resistant Major Depression (TRD).
Brief Title: Efficacy and Safety of Fixed Doses of BMS 820836 in the Treatment of Patients With Treatment Resistant Major Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CN162-007; 2011-000778-71 (EudraCT Number)
Record Dates: First submitted 2011-06-07; First posted 2011-06-08 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-09

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Duloxetine Hydrochloride; Escitalopram; 6-(2-methyl-4-(2-naphthyl)-1,2,3,4-tetrahydroisoquinolin-7-yl)pyridazin-3-amine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Arm 1: Duloxetine / Escitalopram + BMS-820836 placebo (Active Comparator)
  Interventions: Drug: Duloxetine; Drug: Escitalopram; Drug: BMS-820836 Placebo
- Arm 2: BMS-820836 (0.25 mg) + BMS-820836 placebo (Experimental)
  Interventions: Drug: BMS-820836 Placebo; Drug: BMS-820836
- Arm 3: BMS-820836 (0.50 mg) + BMS-820836 placebo (Experimental)
  Interventions: Drug: BMS-820836 Placebo; Drug: BMS-820836
- Arm 4: BMS-820836 (1.0 mg) + BMS-820836 placebo (Experimental)
  Interventions: Drug: BMS-820836 Placebo; Drug: BMS-820836
- Arm 5: BMS-820836 (2.0 mg) + BMS-820836 placebo (Experimental)
  Interventions: Drug: BMS-820836 Placebo; Drug: BMS-820836

INTERVENTIONS:
Drug: Duloxetine — Capsule, Oral, 30-60mg/day, once daily, 7 weeks (Phase B), 7weeks (Phase C&D)
  Other Names: Cymbalta
  Arms: Arm 1: Duloxetine / Escitalopram + BMS-820836 placebo
Drug: Escitalopram — Capsule, Oral, 10-20 mg/day, once daily, 7 weeks (Phase B), 7 weeks (Phase C&D)
  Other Names: Lexapro
  Arms: Arm 1: Duloxetine / Escitalopram + BMS-820836 placebo
Drug: BMS-820836 Placebo — Tablet, Oral, 0.0mg, once daily, 13 weeks (Phase B&C)
Drug: BMS-820836 — Tablet, Oral, 0.25mg, once daily, 6 weeks (Phase C)
  Arms: Arm 2: BMS-820836 (0.25 mg) + BMS-820836 placebo
Drug: BMS-820836 — Tablet, Oral, 0.5 mg, once daily, 6 weeks (Phase C)
  Arms: Arm 3: BMS-820836 (0.50 mg) + BMS-820836 placebo
Drug: BMS-820836 — Tablet, Oral, 1.0 mg, once daily, 6 weeks (Phase C)
  Arms: Arm 4: BMS-820836 (1.0 mg) + BMS-820836 placebo
Drug: BMS-820836 — Tablet, Oral, 2.0 mg, once daily, 6 weeks (Phase C)
  Arms: Arm 5: BMS-820836 (2.0 mg) + BMS-820836 placebo

SUMMARY:
The purpose of the study is to evaluate the efficacy of study drug (BMS-820836) as compared with continued Duloxetine/Escitalopram in the treatment of patients with treatment resistant depression (TRD).

ELIGIBILITY:
Inclusion Criteria:

* Men and women of age 18-65 years (Argentina minimum age will be 24 years of age)
* Patients must be able to understand the nature of the study, agree to comply with the prescribed dosage regimens, report for regularly scheduled office visits, and communicate to study personnel about adverse events and concomitant medication use.
* Patients with a diagnosis of Major Depressive Disorder, currently experiencing a Major Depressive Episode, as defined by Diagnostic and Statistical Manual of Mental Disorders- Fourth Edition (Text Revision)[DSM IV TR] criteria. The current depressive episode must be > 8 weeks in duration and < 3 years duration.
* In the current Major depressive disorder (MDD) episode, patients should report a history of inadequate response to 1-3 adequate trials of antidepressant treatment.
* Patients must have a 17-item Hamilton Depression Rating Scale (HAM-D17) total score ≥ 18 at Screening and Baseline.

Exclusion Criteria:

* Patients who report an inadequate response (less than 50% reduction in depressive symptom severity) to more than three adequate trials of antidepressant treatments during the current depressive episode.
* Patients who have failed Duloxetine and Escitalopram at an adequate dose and for an adequate duration in their current episode.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 976 (Actual)
Dates: Start 2011-07; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline to endpoint in the Montgomery Asberg Depression Rating Scale (MADRS) total score | Week 13

SECONDARY OUTCOMES:
Change from baseline to endpoint in mean Sheehan Disability Scale (SDS) score. | Week 13

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (86):
- United States (48):
  - Birmingham Psychiatry Pharmaceutical Studies, Inc., Birmingham, Alabama
  - Arkansas Psychiatric Clinic Clinical Research Trials, P.A., Little Rock, Arkansas
  - Catalina Research Institute, Llc, Chino, California
  - Behavioral Research Specialists, Llc, Glendale, California
  - Pacific Clinical Research Medical Group, Orange, California
  - Anderson Clinical Research, Redlands, California
  - Affiliated Research Institute, San Diego, California
  - Artemis Institute For Clinical Research, San Diego, California
  - Sharp Mesa Vista Hospital, San Diego, California
  - Western Affiliated Research Institute, Denver, Colorado
  - Connecticut Clinical Research, Cromwell, Connecticut
  - Meridien Research, Brooksville, Florida
  - Gulfcoast Clinical Research Center, Fort Myers, Florida
  - Amit Vijapura, Jacksonville, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Janus Center For Psychiatric Research, West Palm Beach, Florida
  - Emory University, Atlanta, Georgia
  - Uptown Research Institute, Llc, Chicago, Illinois
  - Clinco, Terre Haute, Indiana
  - Clinical Trials Technology, Inc, Prairie Village, Kansas
  - Ert, Shreveport, Louisiana
  - Mclean Hospital, Belmont, Massachusetts
  - Bio Behavioral Health, Toms River, New Jersey
  - Albuquerque Neuroscience, Inc., Albuquerque, New Mexico
  - Comprehensive Clinical Development, Inc, Fresh Meadows, New York
  - Bioscience Research, Llc, Mount Kisco, New York
  - Village Clinical Research, Inc., New York, New York
  - Northcoast Clinical Trials, Inc, Beachwood, Ohio
  - Patient Priority Clinical Sites, Llc, Cincinnati, Ohio
  - Neurology & Neuroscience Center Of Ohio, Toledo, Ohio
  - Suburban Research Associates, Media, Pennsylvania
  - Keystone Clinical Studies, Llc, Norristown, Pennsylvania
  - Ert, Pittsburgh, Pennsylvania
  - Neuropsychiatric Research Center Of Orange County, Pittsburgh, Pennsylvania
  - Northwest Clinical Research Center, Pittsburgh, Pennsylvania
  - Lincoln Research, Lincoln, Rhode Island
  - Future Search Trials, Austin, Texas
  - Futuresearch Trials Of Dallas, Dallas, Texas
  - Insite Clinical Research, DeSoto, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Grayline Clinical Drug Trials, Wichita Falls, Texas
  - Ericksen Research And Development, Clinton, Utah
  - Clinical Methods Llc, Murray, Utah
  - Neuropsychiatric Associates, Woodstock, Vermont
  - Neuroscience, Inc, Herndon, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Summit Research Network (Seattle) Llc, Seattle, Washington
  - Dean Foundation For Health Research & Education, Middleton, Wisconsin
- Argentina (4):
  - Local Institution, Caba, Buenos Aires
  - Local Institution, La Plata, Buenos Aires
  - Local Institution, Córdoba, Córdoba Province
  - Local Institution, Mendoza, Mendoza Province
- Australia (4):
  - Local Institution, Brisbane, Queensland
  - Local Institution, Adelaide, South Australia
  - Local Institution, Heidelberg, Victoria
  - Local Institution, Nedlands, Western Australia
- Local Institution, Vienna, Austria
- Canada (5):
  - Local Institution, Vancouver, British Columbia
  - Local Institution, Bathurst, New Brunswick
  - Local Institution, Ottawa, Ontario
  - Local Institution, Toronto, Ontario
  - Local Institution, Montreal, Quebec
- France (5):
  - Local Institution, Montpellier, France
  - Local Institution, Dole
  - Local Institution, Douai
  - Local Institution, Élancourt
  - Local Institution, Jonzac
- India (9):
  - Local Institution, Tirupati, Andhra Pradesh
  - Local Institution, Visakhapatnam, Andhra Pradesh
  - Local Institution, Ahmedabad, Gujarat
  - Local Institution, Mumbai, Maharashtra
  - Local Institution, Pune, Maharashtra
  - Local Institution, Lucknow, Uttar Pradesh
  - Local Institution, Chennai
  - Local Institution, Pune
  - Local Institution, Varanasi
- Italy (3):
  - Local Institution, Pisa
  - Local Institution, Roma
  - Local Institution, Siena
- Local Institution, Ponce, Puerto Rico
- South Africa (2):
  - Local Institution, Pretoria, Gauteng
  - Local Institution, Durban, KwaZulu-Natal
- Local Institution, Barcelona, Spain
- United Kingdom (3):
  - Local Institution, London, Greater London
  - Local Institution, Edgware, Middlesex
  - Local Institution, Birmingham, West Midlands

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx